CLINICAL TRIAL: NCT05701345
Title: Prospective, Multicenter, Assessor-blind, Randomized, Comparative, Pivotal Study to Evaluate the Efficacy and Safety of Wearable Visual Device (HMD)-VR-based Software Medical Device(OMNIFIT DTx-MDD) for Patients with Depressive Disorder
Brief Title: Study of Virtual Reality-based Medical Device for Patients with Depressive Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Omni C&S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OMNI_MDD_01
Record Dates: First submitted 2023-01-12; First posted 2023-01-27 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-11

CONDITIONS: Depressive Disorder; Major Depressive Disorder; Depressive Episode
Keywords: mild and moderate depressive disorder
MeSH Terms: conditions — Depressive Disorder; Depressive Disorder, Major; Lymphoma, Follicular | interventions — Antidepressive Agents

STUDY DESIGN:
Intervention Model Description: Multiple-Group Assignment
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- medical device used group (Experimental): Wearable visual device(HMD)-VR-based software medical device(OMNIFIT DTx-MDD)
  Interventions: Device: OMNIFIT DTx-MDD; Other: standard treatment
- medical device unused group (Placebo Comparator): Patients receiving only standard treatment
  Interventions: Other: standard treatment

INTERVENTIONS:
Device: OMNIFIT DTx-MDD — This software medical device consists of multifaceted interventions (breathing training, cognitive rehabilitation training, binaural beat training, concentration training) that help improve depressive disorder, and is automatically executed for 35 minutes per session
  Other Names: Wearable visual device-based software medical device
  Arms: medical device used group
Other: standard treatment — It is based on the Korean Medical Association's clinical treatment guidelines for depression or the Korean Medical Association's Korean Medical Association/Korean Depression Management Association's 2021 guidelines for drug treatment for depression disorders.
  Standard treatment will be performed according to the judgment of the attending physician reflecting the clinical situation based on these treatment guidelines.
  Other Names: Antidepressant

SUMMARY:
This study apply a wearable visual device (HMD)-VR-based software medical device for patients with depressive disorder for 8 weeks.

The investigator would like to confirm evaluate the safety and efficacy of the wearable visual device(HMD)-VR-based software medical device effect of improving depressive disorder in patients.

DETAILED DESCRIPTION:
Trial subject is a mild and moderate patients diagnosed with depressive disorder The test group is a wearable visual device(HMD)-VR-based software medical device(OMNIFIT DTx-MDD) and patients who have received standard treatment.

The number of subjects is 162(Two groups, 81 people per group, 15% dropout rate included) Participating institutions are five including Catholic University of Korea Seoul ST.

The clinical trial method is as follows. Subjects who are satisfied with all selection/exclusion criteria and agree to participate in clinical trials are classified into groups that combine test software medical devices and standard treatment based on Visit 2 (Baseline) and groups that perform simple standard treatment. After that, necessary tests are performed at 2, 4, 6, and 8 weeks, and changes in depressive disorder and depressive disorder evaluation scale are confirmed, and safety is evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. right-handed men and women
2. If you agree to participate in this clinical trial and voluntarily sign a written consent form
3. If you can understand and cooperate with the contents of this clinical trial
4. If you have a wireless internet(Wifi) environment
5. Diagnosed by a psychiatrist as major depressive disorder according to the Diagnostic and Statistical Manual of Mental Disorder 5th edition(DSM-5) or other specified depressive disorder
6. Mild or moderate depressive episodes with a total hdrs score of 7 or more and 24 or less
7. If there was no change in the type and dose of antidepressants and antipsychotics taken within 4 weeks prior to participation in this clinical trial

Exclusion Criteria:

1. if you are pregnant
2. Schizophrenia, schizoaffective disorder, schizophrenic disorder, or a psychotic disorder not otherwise classified or diagnosed in the past
3. If you have current bipolar disorder or have been diagnosed with bipolar disorder in your past history
4. Accompanied by organic mental disorder, epilepsy/convulsive disorder
5. Current eating disorders, alcohol and other substance-related disorders, and obsessive-compulsive disorder
6. Uncontrolled and unstable clinically significant physical condition
7. In cases where psychiatric evaluation and maintenance of treatment are difficult due to other serious acute physical illnesses
8. If you have received electroconvulsive therapy and transcranial magnetic stimulation therapy for a current depressive episode
9. Treatment-resistant depressive disorder for which there was no effect even after using two or more antidepressants in sufficient doses and for a sufficient period of time (6 weeks) for the current depressive episode
10. Currently requiring inpatient treatment for a psychiatric disorder other than depressive disorder (ex. alcohol dependence, substance abuse)
11. If the risk of suicide, self-harm, or other harm is judged to be high according to the evaluation of the study director
12. Current depressive episode accompanied by psychotic symptoms
13. Cases in which a therapeutic intervention for a clinical trial cannot be performed due to deterioration of eyesight or hearing
14. Current treatment with mood stabilizers (lithium, valproate, carbamazepine, lamotrigine) for depressive episodes
15. Those who are unable to participate in clinical trials due to the judgment of other researchers
16. Those who cannot read the consent form (ex. illiterate, foreigners)

Ages: 19 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 162 (Actual)
Dates: Start 2023-03-09 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Comparison of change in Hamilton Depression Rating Scale total score | 8 weeks
  The comparison of changes in Hamilton Depression Rating Scale total score between each group is evaluated by Student t-test performing two independent samples.
  The minimum value is 0 points and the maximum value is 52 points, with higher scores indicating more severe depressive symptoms.

SECONDARY OUTCOMES:
Comparison of response rate and remission rate by Hamilton Depression Rating Scale | 8 weeks
  chi-squared test or Fisher's exact test is performed to compare response rates (reduction of 50% or more from baseline) and remission rates (Hamilton Depression Rating Scale total score of 6 points or less) by Hamilton Depression Rating Scale between and within groups, and the within-group comparison is based on the frequency of improvement. Evaluate by performing McNemar test for The minimum value is 0 points and the maximum value is 52 points, with higher scores indicating more severe depressive symptoms.
Comparison of Changes in Patient Health Questionnaire-9 Scores | 8 weeks
  The comparison of changes in the Patient Health Questionnaire-9 score between each group is performed by an independent two-sample student t-test, and the comparison within groups is evaluated by a paired-sample t-test.
  The Patient Health Questionnaire-9 score has a minimum value of 0 and a maximum value of 27 points, with higher scores indicating more severe depression.
Comparison of Changes in Clinical Global Impression - Severity & Clinical Global Impression | 8 weeks
  The comparison of changes in the Clinical Global Impression - Severity & Clinical Global Impression - Improvement scores between each group is performed by an independent two-sample student t-test, and the comparison within groups is evaluated by a paired-sample t-test.
  The Clinical Global Impression - Severity & Clinical Global Impression has a minimum value of 0 and a maximum value of 7 points, with higher scores indicating more severe depression.
Comparison of side effects | 8 weeks
  Comparison of side effects between each group is evaluated by performing a chi-squared test or Fisher's exact test after using the test software medical device.
Comparison of adverse events | 8 weeks
  Comparison of side adverse events each group is evaluated by performing a chi-squared test or Fisher's exact test after using the test software medical device.
Comparison of dropout rates | 8 weeks
  Comparison of dropout rates events each group is evaluated by performing a chi-squared test or Fisher's exact test after using the test software medical device.

CONTACTS AND LOCATIONS:
Overall Officials: Youngsup Woo, Principal Investigator — Yeouido St. Mary's Hospital
Locations (5):
- South Korea (5):
  - Inje University Ilsan Palk Hospital, Ilsan
  - Jeju National University Hospital, Jeju City
  - Seoul ST. Mary's Hospital, Seoul
  - Yeouido ST. Mary's Hospital, Seoul
  - ST. Vincent's Hospital, Suwon